CLINICAL TRIAL: NCT04025229
Title: Pre-operative Window Study of Interval Exercise Training as a Therapy for Endometrial Cancer
Brief Title: High Intensity Interval Training in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC 1839; 1R21CA235029-01 (NIH)
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will complete HIIT training prior to surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT exercise (Experimental): Participants will perform HIIT exercises as instructed by the study team in the weeks prior to standard of care surgery
  Interventions: Behavioral: HIIT exercise

INTERVENTIONS:
Behavioral: HIIT exercise — High intensity interval training (4 to 6 sessions) prior to surgery

SUMMARY:
This interventional trial recruits women with endometrial cancer to participate in high intensity interval training (HIIT) prior to their standard of care surgery. The study will evaluate tissue and blood to determine if HIIT training has anti-cancer effects. P

DETAILED DESCRIPTION:
Primary Objectives:

1. Determine the anti-proliferative effect of HIIT on the endometrium of women with endometrial cancer 2. Participants will undergo baseline testing, be taught how to perform personalized HIIT training prior to surgery, and repeat testing after surgery. Tissue specimens will be collected from standard of care biopsy (no extra biopsy needed) and during surgery. Blood will be collected twice during standard of care blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of endometrial cancer who are to undergo hysterectomy and staging
* Between 40-75 years old
* Body mass index of 30-50 kg/m2
* Endometrioid histology endometrial cancer
* Presumed clinically early stage disease (disease confined to uterus only)
* Have access to a Smart Phone
* Have access to email
* Agree to visit the exercise and sport science laboratory within 2 days of SOC visit for baseline testing if enrollment procedures cannot be done on the same day.

Agree to visit clinic 2 (+/-2wks) weeks after surgery for SOC follow-up and post surgery visit, or willing to return to exercise and sport science laboratory 2 (+/-2wks) weeks post-surgery

Exclusion Criteria:

* Meets American College of Sports Medicine Guidelines for physical activity (150 minutes / week)
* Currently doing HIIT
* Hospitalization for a stroke, heart attack, or heart failure, or had surgery for blocked arteries in the past 3 months
* Active diagnosis of psychosis or current uncontrolled substance abuse disorder
* Insulin-dependent diabetes
* Currently in another EC intervention
* Severe dementia or other memory loss condition
* Severe mental health disorder
* Severely impaired hearing or speech
* Inability to speak English
* Musculoskeletal or neuromuscular condition that limits physical activity Any condition, in the opinion of the investigators, which would prohibit safe participation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study recruits women with endometrial cancer
Enrollment: 30 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled were enrolled at a single North Carolina site between 09/23/2019 and 09/08/2022.
Pre-assignment Details: Thirty participants consented and began the study.
Groups:
- Control Arm: No HIIT exercise prior to surgery
- HIIT Exercise: Participants will perform HIIT exercises as instructed by the study team in the weeks prior to standard of care surgery.
  HIIT exercise: High-intensity interval training (4 to 6 sessions) prior to surgery.
Period: Overall Study
Arm/Group | Control Arm | HIIT Exercise
Started | 10 | 20
Completed | 9 | 16
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | HIIT Exercise | Total
Number analyzed (Participants) | 9 | 16 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (5.3) | 54.9 (8.2) | 56.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 15 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Proliferative Markers in Endometrium Before and After HIIT Exercises
Description: Change in Ki-67 proliferation values within the HIIT intervention group between the initial biopsy and the surgical biopsy. The percentage of tumor cells that are positive for Ki-67, indicating they are in the active phases of the cell cycle (not resting). Low Ki-67 (<10-15%): Slower-growing tumor. Intermediate (15-30%): Moderately proliferative. High (>30%): Fast-growing, potentially more aggressive.
Time Frame: 3 years
Population: Participants who started the study and provided a sample were included.
Measure: Mean (Standard Deviation); unit: Percentage of cells expressing Ki67
Groups:
- Control Arm- Baseline: The sample provided by participants who will perform HIIT exercises as instructed by the study team in the weeks prior to standard of care surgery at baseline.
- Control Arm -At Surgery: The sample provided by participants who will perform HIIT exercises as instructed by the study team in the weeks prior to standard of care surgery at surgery.
- HIIT- Baseline: The sample provided by participants who will perform HIIT exercises as instructed by the study team at baseline.
- HIIT -At Surgery: The sample provided by participants who will perform HIIT exercises as instructed by the study team during surgery.
Arm/Group | Control Arm- Baseline | Control Arm -At Surgery | HIIT- Baseline | HIIT -At Surgery
Number analyzed (Participants) | 8 | 8 | 16 | 16
Percentage of cells expressing Ki67 | 21.7 (12.2) | 15.1 (14.4) | 21.7 (12.2) | 20.2 (15.7)

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment.
Description: The protocol did not require adverse event (AE) assessment; therefore, AE data were not systematically collected. However, if participants reported discontinuation from the study due to an adverse event or death, these were recorded as non-specific events.
Arm/Group | HIIT Exercise
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04025229/Prot_SAP_000.pdf